CLINICAL TRIAL: NCT05954221
Title: Red Cell Lysis Buffer Application Versus Conventional Sample Processing in Endoscopic Ultrasonography (EUS)-Guided Biopsy for Solid Pancreatic Lesions
Brief Title: Red Cell Lysis Buffer Application Versus Conventional Sample Processing in EUS-FNB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Department of Gastroenterology, Changhai Hospital, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: RBC lysis buffer
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Pancreatic Diseases
Keywords: EUS-FNB; sample processing; solid pancreatic lesion
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red cell lysis buffer (RCLB) group (Experimental): Patients assigned to this group will receive EUS-FNB as routine. The obtained tissue will be processed with red cell lysis buffer and underwent histological evaluation.
  Interventions: Procedure: Red cell lysis buffer (RCLB) application
- conventional group (Active Comparator): Patients assigned to this group will receive EUS-FNB as routine. The obtained tissue will be fixed with formalin as usual and underwent histological evaluation.
  Interventions: Procedure: Conventional processing

INTERVENTIONS:
Procedure: Red cell lysis buffer (RCLB) application — The tissue is lysed with 50% concentration of RCLB for 15 min on a shaking device. If the lysis is judged to be insufficient, it can be repeated one more time. Finally, the treated tissue will be fixed with 10% formalin.
  Arms: Red cell lysis buffer (RCLB) group
Procedure: Conventional processing — The tissue is fixed with 10% formalin.
  Arms: conventional group

SUMMARY:
The goal of this clinical trial is to evaluate the application of red cell lysis buffer (RCLB) versus conventional sample processing in endoscopic ultrasonography (EUS)-guided biopsy for solid pancreatic lesions. The main questions it aims to answer are:

whether the application of red cell lysis buffer improves histological tissue quality by decreasing blood contamination.

Participants with solid pancreatic lesions who needs histological diagnosis will receive EUS-guided biopsy. The obtained specimens will be processed by RCLB and conventional formalin solution.

Researchers will compare the blood contamination score of specimens in RCLB group with the conventional group see if the blood contamination can be improved.

ELIGIBILITY:
Inclusion Criteria:

18 to 80 years old; Solid pancreatic lesions confirmed by clinical and CT/MRI/ PET imaging. Signed written informed consent

Exclusion Criteria:

Contraindication of EUS-guide procedure or technical infeasibility (e.g.,coagulation disorder, anatomical changes, large vessels along the puncture path) Pregnant Patient is enrolled in any other clinical protocol or investigational trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Microscopic blood contamination assessments | 2 months
  Microscopic blood contamination is assessed by grading the percentage of the area of the blood cells in the entire ×40 field of view (score 3, < 25 %; score 2, 25 % - 50%; score 1, > 50 %; score 0, no material)

SECONDARY OUTCOMES:
Tissue integrity assessments | 2 months
  The tissue integrity on histological analysis was also graded into 3 levels: Grade A, existing core tissue (defined as an architecturally intact piece of tissue with a long axis measuring at least 550 μm), which can clearly characterize the lesion, and is sufficient for diagnosis; Grade B, existing core fragments, which does not meet the criteria for architecturally intact histology, but can still yield a diagnosis based on cell morphology; and Grade C, no lesion tissue found, and a diagnosis cannot be made based on the sample.
Macroscopic blood contamination assessments | 2 months
  Macroscopic visual quality of histopathological samples is assessed by grading the percentage of red (blood) component ejected from the needle on a glass slide (score 4, white tissue only; score 3, < 25 %; score 2, 25 % - 50%; score 1, > 50 %; score 0, no material).
Length of white core tissue | 2 months
  MVC (macroscopically visible core), defined as a measurable whitish sample. After collecting the MVCs scattered in the samples, the samples were aligned using a needle, and their length was measured using a ruler.
Diagnostic sensitivity | 2 months
  Diagnostic sensitivity was calculated as the proportion of true positive in patient cases.
Diagnostic accuracy | 2 months
  Diagnostic accuracy was calculated as the proportion of true positive and true negative in all evaluated cases
Diagnostic specificity | 2 months
  Diagnostic specificity were calculated as proportion of true negative in healthy cases
Immunohistochemical assessment | 2 months
  Immunohistochemical assessment: a. Detect whether the expression of membrane proteins is the same in treated and untreated specimens from the additional 3 groups of patients. b. Grading the percentage of the area of non-specific staining of erythrocytes in the entire ×40 field of view. Score of 3, non-specific staining present in < 25% of slides; score of 2, non-specific staining present in 25% - 50% of slides; score of 1, non-specific staining is present in > - 50% of slides
RNA and DNA adequancy | 2 months
  Compare the percentage of samples with sufficient RNA and DNA that could be extracted from.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Shen Li, M.D, Principal Investigator — Department of Gastroenterology, Changhai Hospital, Naval Medical University (Second Military Medical University), Shanghai, China.
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No